CLINICAL TRIAL: NCT05664490
Title: Youth Friendship Bench SA: Optimization of the Friendship Bench Mental Health Intervention for Adolescent Girls and Young Women in South African PrEP Delivery Settings
Brief Title: Friendship Bench Mental Health Intervention for Adolescent Girls and Young Women in South African PrEP Delivery Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37680; 4R00MH123369-03 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Depression; Pre-Exposure Prophylaxis
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-Care Mental Health Services (No Intervention): Participants randomized to this group will receive standard-of-care mental health services as specified in the South African Department of Health Adult Primary Care Guidelines.
- Youth Friendship Bench SA + Standard-of-Care (Experimental): Participants randomized to this group will receive the Youth Friendship Bench SA intervention in addition to standard-of-care mental health services as specified in the South African Department of Health Adult Primary Care Guidelines.
  Interventions: Behavioral: Youth Friendship Bench SA

INTERVENTIONS:
Behavioral: Youth Friendship Bench SA — The intervention includes: 5 individual counseling sessions; one optional in-person or WhatsApp-based group counseling session; optional remote counseling sessions; and optional one-way SMS messages to provide reminders about upcoming visits. During the initial session, participants will meet with the trained counselor to discuss mental health challenges, identify problems in their life that affect their mental health and PrEP use, generate alternative solutions, make decisions about the alternatives, and collaboratively decide on a plan to implement the solutions. During follow-up counseling sessions, participants will discuss progress in implementing solutions to address the problems they identified in prior sessions with the lay counselor. They will also discuss any other mental health challenges and problems in their life that affect their mental health and PrEP use which they would like to address.
  Arms: Youth Friendship Bench SA + Standard-of-Care

SUMMARY:
Adolescent girls and young women (AGYW) at risk of HIV in sub-Saharan Africa, frequently (20-50%) have symptoms of common mental disorders, including depression, anxiety, and stress. These symptoms are associated with suboptimal adherence to HIV pre-exposure prophylaxis (PrEP), a highly effective HIV prevention approach. In this project, the team seeks to address poor mental health and consequent impacts on PrEP adherence and among AGYW at risk of HIV by testing an evidence-based mental health intervention (the Youth Friendship Bench SA) adapted for PrEP delivery programs.

DETAILED DESCRIPTION:
This is a randomized hybrid implementation-effectiveness trial which will be conducted in a real-world healthcare setting. Eligible women who accept open-label daily oral PrEP (n=110) will be enrolled and randomized to either the Youth Friendship Bench SA intervention (plus standard-of-care mental health services as needed) or standard-of-care mental health services alone. Randomization will be conducted in a 1:1 ratio with randomly-sized blocks of ≤10.

HIV-uninfected women ages 18-25 in Johannesburg, South Africa, who have symptoms of common mental disorders as evidenced by a score greater than or equal to 7 on the SRQ-20 will be eligible to enroll.

The investigators hypothesize that the Youth Friendship Bench SA will significantly improve PrEP adherence and reduce symptoms of common mental disorders among AGYW at Month 3.

ELIGIBILITY:
Inclusion Criteria:

* Female 18-25 years of age at screening
* Documentation of symptoms of a common mental disorder, as evidenced by a score greater than or equal to 7 on the Self Reporting Questionnaire 20-item (SRQ-20)
* Willingness to enroll and be randomized to either the Youth Friendship Bench SA or standard-of-care mental health services
* Written informed consent (obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study.
* Able to verbally communicate in one or more study languages to ensure participation in the counseling sessions (English, isiZulu)
* Taking PrEP at the Ward 21 clinic, as determined by clinic records. PrEP provision will be conducted by the clinic following National PrEP Guidelines and will not be part of study-specific procedures.

Exclusion Criteria:

* Not on PrEP and/or not intending to use PrEP for the duration of the study
* Planning to relocate in the next three months
* Report of suicidal intent or self harm
* Active, unmanaged mental health disorders, including untreated or severe somatic symptoms and active psychiatric symptoms (e.g., hallucinations)
* Reactive or positive HIV test at enrollment (based on clinic records only; HIV testing will not be performed under this protocol)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Velloza, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Wits Reproductive Health Institute, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be available at the end of the project by contacting the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: End of study.
Access Criteria: Reasonable request to the Principal Investigator.

REFERENCES:
- [Background] Velloza J, Hosek S, Donnell D, Anderson PL, Chirenje M, Mgodi N, Bekker LG, Delany-Moretlwe S, Celum C; HPTN 082 study group. Assessing longitudinal patterns of depressive symptoms and the influence of symptom trajectories on HIV pre-exposure prophylaxis adherence among adolescent girls in the HPTN 082 randomized controlled trial. J Int AIDS Soc. 2021 Jun;24 Suppl 2(Suppl 2):e25731. doi: 10.1002/jia2.25731. PMID 34164929
- [Background] Remien RH, Stirratt MJ, Nguyen N, Robbins RN, Pala AN, Mellins CA. Mental health and HIV/AIDS: the need for an integrated response. AIDS. 2019 Jul 15;33(9):1411-1420. doi: 10.1097/QAD.0000000000002227. PMID 30950883
- [Background] Abas M, Nyamayaro P, Bere T, Saruchera E, Mothobi N, Simms V, Mangezi W, Macpherson K, Croome N, Magidson J, Makadzange A, Safren S, Chibanda D, O'Cleirigh C. Feasibility and Acceptability of a Task-Shifted Intervention to Enhance Adherence to HIV Medication and Improve Depression in People Living with HIV in Zimbabwe, a Low Income Country in Sub-Saharan Africa. AIDS Behav. 2018 Jan;22(1):86-101. doi: 10.1007/s10461-016-1659-4. PMID 28063075
- [Background] Chibanda D, Weiss HA, Verhey R, Simms V, Munjoma R, Rusakaniko S, Chingono A, Munetsi E, Bere T, Manda E, Abas M, Araya R. Effect of a Primary Care-Based Psychological Intervention on Symptoms of Common Mental Disorders in Zimbabwe: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2618-2626. doi: 10.1001/jama.2016.19102. PMID 28027368
- [Background] Udedi M, Stockton MA, Kulisewa K, Hosseinipour MC, Gaynes BN, Mphonda SM, Mwagomba BM, Mazenga AC, Pence BW. Integrating depression management into HIV primary care in central Malawi: the implementation of a pilot capacity building program. BMC Health Serv Res. 2018 Jul 31;18(1):593. doi: 10.1186/s12913-018-3388-z. PMID 30064418
- [Background] Brooks MJ, Phetogo BK, Schwennesen H, Phoi O, Tshume O, Matshaba M, Lowenthal E. Building a Community Based Mental Health Program for Adolescents in Botswana: Stakeholder Feedback. Community Ment Health J. 2022 Aug;58(6):1068-1075. doi: 10.1007/s10597-021-00915-5. Epub 2021 Nov 26. PMID 34826035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on referral from clinic personnel during clinic visits between April and October of 2023. The first participant was enrolled in April 2023 and the last participant was enrolled in October 2023.
Pre-assignment Details: 222 participants were assessed for eligibility. 93 did not meet eligibility criteria and thus were excluded from randomization. 3 screened participants declined participation and 10 participants did not complete enrollment procedures. 116 participants were randomized.
  We enrolled 6 additional participants, over our target sample size of 110 participants, to replace 6 participants who terminated the study early (6 had terminated within 4 weeks, at the time of enrollment close).
Groups:
- Standard-of-Care Mental Health Services: Participants randomized to this group will receive standard-of-care mental health services as specified in the South African Department of Health Adult Primary Care Guidelines. Participants randomized to this group will return for visits at Weeks 4 and 12.
- Youth Friendship Bench SA + Standard-of-Care: Participants randomized to this group will receive the Youth Friendship Bench SA intervention in addition to standard-of-care mental health services as specified in the South African Department of Health Adult Primary Care Guidelines. Participants randomized to this group will receive counseling at Enrollment, Weeks 2, 4, 8, and 12.
Period: Overall Study
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Started | 58 | 58
Week 2 | 58 | 57
Week 4 | 41 | 35
Week 8 | 41 | 37
Week 12 | 44 | 36
Completed | 44 | 35
Not Completed | 14 | 23
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 14 | 22

BASELINE CHARACTERISTICS:
Population: One Youth Friendship Bench SA + Standard-of-Care participant was randomized but did not complete enrollment surveys and thus is excluded from Baseline Characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 21 [20 to 23] | 21 [19 to 22] | 21 [20 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
SRQ-20 Score [Median (Inter-Quartile Range); unit: Score] — The SRQ-20 is a validated measure to detect non-specific psychological distress with possible values between 0 and 20. A higher score indicates more depressive symptoms.
  Score | 8 [7 to 10] | 9 [8 to 10] | 9 [7 to 10]
PHQ-9 [Median (Inter-Quartile Range); unit: Score] — The PHQ-9 is a validated scale to measure depressive symptoms. It has a possible range of 0-27. Higher scores indicate more depressive symptoms.
  Score | 8.5 [6.3 to 11] | 8 [5 to 12] | 8 [5.5 to 11.5]
GAD-7 [Median (Inter-Quartile Range); unit: Score] — The GAD-7 is a validated scale to measure anxiety symptoms. It has a possible range of 0-21. A higher score indicates more anxiety symptoms.
  Score | 6 [4.3 to 10] | 7 [5 to 11] | 6 [4.5 to 10]
Has experienced gender-based violence [Count of Participants; unit: Participants] — Gender-based violence questions based on the World Health Organization's screening tool.
  Participants | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: PrEP Adherence at Week 12
Description: The proportion of participants with PrEP adherence at Month 3, defined as tenofovir (TFV) concentrations ≥1500 ng/mL in urine measured using a urine POC assay
Time Frame: Week 12
Population: This data is from an intent-to-treat analysis that included all randomized participants that completed enrollment procedures (N = 115). We used multiple imputation using chained equations (MICE) to account for missingness due to missed visits and early terminations. Randomly imputed values were generated from 100 imputations and, to meet assumptions that data were conditionally missing at random, we included baseline variables associated with missingness in our imputation model.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 58 | 57
Participants | 29 | 22
Statistical Analysis 1: Comparison: Standard-of-Care Mental Health Services; Test type: Superiority; p = 0.44, Poisson regression — The threshold for statistical significance is 0.05; We used Poisson regression with a log-link and robust standard errors to assess the effect of our intervention on PrEP adherence at Week 12; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.64 to 1.22] — The Standard of Care Mental Health Services arm was the reference category for the risk ratio

2. Primary Outcome: Change in Proportion of Participants With Self Reporting Questionnaire 20-Item (SRQ-20) Scores Below 7
Description: The change in the proportion of participants with SRQ-20 scores <7 will be reported. Mental health symptoms will be measured on the SRQ-20, with a score below 7 indicating no or mild symptoms of depression, anxiety, or stress. SRQ-20 scores are calculated as the sum of responses across 20 items asking about symptoms of common mental disorders (e.g. depression, anxiety). Each item has a yes or no response and 'yes' responses are coded as '1' and 'no' responses are coded as '0' (possible score range = 0-20, with higher scores indicating greater severity of common mental disorder symptoms).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 58 | 57
Participants | 29 | 23
Statistical Analysis 1: Comparison: Standard-of-Care Mental Health Services; Test type: Superiority; p = 0.99, Poisson regression — The threshold for statistical significance was 0.05; We used Poisson regression with a log-link and robust standard errors to assess the effect of our intervention on reduced CMD symptoms at Week 12; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.71 to 1.42] — The reference category for the risk ratio presented is the Standard of Care Mental Health Services arm

3. Secondary Outcome: PrEP Adherence at Week 4
Description: The proportion of participants with PrEP adherence at Week 4, defined as tenofovir (TFV) concentrations ≥1500 ng/mL in urine measured using a urine POC assay
Time Frame: Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 58 | 57
Participants | 25 | 29
Statistical Analysis 1: Comparison: Standard-of-Care Mental Health Services; Test type: Superiority; p = 0.03, Poisson regression — The threshold for statistical significance was 0.05; We used Poisson regression with a log-link to estimate to assess the effect of our intervention on PrEP adherence at Week 4; Risk Ratio (RR) = 1.40, 95% CI 2-sided [1.03 to 1.89] — The Standard of Care Mental Health Services arm was the reference category for the risk ratio

4. Secondary Outcome: Change in Proportion of Participants With Self Reporting Questionnaire 20-Item (SRQ-20) Scores Below 7
Description: as for outcome 2
Time Frame: Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 58 | 57
Participants | 20 | 15
Statistical Analysis 1: Comparison: Standard-of-Care Mental Health Services; Test type: Superiority; p = 0.37, Poisson regression — The threshold for statistical significance was 0.05; We used Poisson regression with a log-link to assess the effect of the intervention on common mental disorders at Week 4; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.50 to 1.29] — The Standard of Care Mental Health Services arm was the reference category

5. Secondary Outcome: Acceptability of Youth Friendship Bench SA
Description: Acceptability of the Youth Friendship Bench SA intervention as measured by the 4-item Acceptability of Intervention Measure (AIM). The AIM used in this study consists of 4 questions with scales values that range from 1 to 4. Higher scores indicate greater acceptability.
Time Frame: 12 Weeks
Population: The acceptability of the Youth Friendship Bench SA intervention was only asked among Youth Friendship Bench SA + Standard of Care participants who attended the week 12 visit (n = 35).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 0 | 35
score on a scale |  | 3.5 [3.0 to 4.0]

6. Secondary Outcome: Feasibility of Youth Friendship Bench SA
Description: Feasibility of the Youth Friendship Bench SA intervention as measured by the 4-item Feasibility of Intervention Measure (FIM). The FIM used in this study consists of 4 questions with scales values that range from 1 to 4. Higher scores indicate greater acceptability.
Time Frame: 12 Weeks
Population: The feasibility of the Youth Friendship Bench SA intervention was only asked among Youth Friendship Bench SA + Standard of Care participants who attended the week 12 visit (n = 35).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 0 | 35
score on a scale |  | 3.75 [3.25 to 4.0]

7. Secondary Outcome: Appropriateness of Youth Friendship Bench SA
Description: Appropriateness of the Youth Friendship Bench SA intervention as measured by the 4-item Intervention Appropriateness Measure (IAM). The IAM used in this study consists of 4 questions with scales values that range from 1 to 4. Higher scores indicate greater acceptability.
Time Frame: 12 Weeks
Population: The appropriateness of the Youth Friendship Bench SA intervention was only asked among Youth Friendship Bench SA + Standard of Care participants who attended the week 12 visit (n = 35).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
Number analyzed (Participants) | 0 | 35
score on a scale |  | 3.25 [3.0 to 4.0]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse Events were non-systematically reported via a REDCap case report form (CRF) for each participant. The CRF did not have to be completed for each participant, and was only completed is an adverse event was reported or discovered.
Arm/Group | Standard-of-Care Mental Health Services | Youth Friendship Bench SA + Standard-of-Care
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/57
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-of-Care Mental Health Services (N=58) | Youth Friendship Bench SA + Standard-of-Care (N=57)
Poison Ingestion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — One Youth Friendship Bench SA + Standard-of-Care participant accidentally ingested rat poison. She was hospitalized. Her counseling sessions showed progress and reduced SRQ-20 scores over time.
Suicidal Attempt (Psychiatric disorders) | 1 (1) | 0 (0) — One Standard of Care Mental Health Services participant deliberately self-harmed and was treated with hospital management and medications.

LIMITATIONS AND CAVEATS:
This study was a pilot study with a small sample size and retention challenges. Retention was lower in the Youth Friendship Bench arm than Standard of Care Mental Health Services arm. We did not collect biomarker data on longer-term PrEP adherence given the short duration of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05664490/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT05664490/SAP_001.pdf